CLINICAL TRIAL: NCT01349933
Title: Multicenter Phase II Study of MK-2206 in Previously Treated Patients With Recurrent and Metastatic Nasopharyngeal Carcinoma
Brief Title: Akt Inhibitor MK2206 in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02581; NCI-2011-02581 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000696863; MC1079 (Other: Mayo Clinic); 8761 (Other: CTEP); P30CA015083 (NIH); N01CM00099 (NIH)
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Recurrent Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx
MeSH Terms: interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Patients receive 200 mg Akt inhibitor MK2206 PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt inhibitor MK2206

INTERVENTIONS:
Drug: Akt inhibitor MK2206 — Given PO
  Other Names: MK2206

SUMMARY:
This phase II trial is studying how well Akt inhibitor MK2206 works in treating patients with recurrent or metastatic head and neck cancer. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients alive and progression-free at 6 months along with the confirmed response rate as a dual primary endpoint..

SECONDARY OBJECTIVES:

I. To evaluate best response and duration of response for patients treated with MK2206 (Akt inhibitor MK2206).

II. To evaluate the overall survival and progression-free survival (PFS) of patients treated with MK2206.

III. To evaluate safety and tolerability of MK2206.

TERTIARY OBJECTIVES:

I. To evaluate the pharmacokinetics of MK2206 in Asian patients. II. To study the pharmacodynamic effect of MK2206 using biomarkers and correlation with cancer-related outcomes.

OUTLINE: This is a multicenter study.

Patients receive Akt inhibitor MK2206 orally (PO) on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection at baseline and periodically during study for pharmacogenomic and pharmacokinetic studies.

After completion of study therapy, patients are followed up for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-keratinizing nasopharyngeal carcinoma that has recurred at locoregional and/or distant sites, and is not amenable to potentially curative radiotherapy or surgery
* Measurable disease according to the RECIST criteria
* Progressed =< 24 months of receiving one or two prior line(s) of chemotherapy for recurrent disease, of which at least one line must contain platinum drugs such as cisplatin, carboplatin or oxaliplatin
* ECOG performance status 0, 1, or 2
* Hemoglobin >= 9 g/dL
* ANC >= 1,500/μL
* Platelet count >= 100,000/μL
* Total bilirubin =< 2.5 times upper limit of normal (ULN)
* ALT =< 2.5 times ULN (=< 5 times ULN for patients with liver metastases)
* Creatinine =< 1.5 times ULN OR creatinine clearance >= 60 mL/min/1.73 m^2
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to donate blood for mandatory correlative research studies
* Negative (serum) pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

Exclusion Criteria:

* Any of the following

  * Chemotherapy =< 4 weeks prior to registration
  * Radiotherapy =< 4 weeks prior to registration
  * Nitrosoureas or Mitomycin C =< 4 weeks prior to registration
  * Those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
  * NOTE: Prior palliative radiotherapy to bone metastases is allowed =< 4 weeks prior to registration
* Prior investigational agents =< 4 weeks prior to registration
* Symptomatic brain metastases; NOTE: primary nasopharyngeal cancers that directly invade the skull base and extend into the infratemporal fossa(e) are not regarded as brain metastases and are not excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 or other agents used in the study
* Prior potent and moderate inhibitors and inducers of CYP3A4 =< 2 weeks prior to registration:

  * Drugs that are forbidden, potent inducers of CYP3A4: phenytoin, phenobarbitone, carbamazepine, barbiturate, rifampicin, St John's Wort.
  * Drugs that significantly affect metabolizing activity by way of enzyme inhibition of CYP3A4: ketoconazole, itraconazole, fluconazole, indinavir, ritonavir, erythromycin, cimetidine, clarithromycin
* Unwillingness to go off other inducers and inhibitors of CYP3A4 during the first 2 cycles of MK-2206; NOTE: avoiding these drugs is critical during the first 2 cycles of MK-2206when blood samples are being taken for the correlative study unless there is an urgent medical need and alternatives are not available
* Poorly controlled diabetes mellitus or insulin controlled diabetes; NOTE: As a general guide, patients with a fasting glucose level > 150 mg/dL (HbA1c <8%, > 8.3 mmol/L), or a random glucose level of >180mg/dL (> 10 mmol/L) is considered to have inadequately controlled diabetes and are not eligible for this study; however, such patients can become eligible in the future if their fasting glucose levels improve with medical treatment
* QTc prolongation (defined as a QTc interval > 450 msec for males and >470 msec for females) or other significant ECG abnormalities; NOTE: patients with clinically significant cardiac conduction abnormalities should be excluded, these include left bundle branch block (LBBB), 2nd or 3rd degree AV block, bifascicular block, sick sinus syndrome, Wolff-Parkinson-white syndrome, sinus bradycardia (< 50bpm); however, patients with asymptomatic right bundle branch block (RBBB) or 1st degree AV block, in the absence of known cardiac disease (e.g. coronary, valvular) are not excluded
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection,
  * Symptomatic congestive heart failure,
  * Unstable angina pectoris,
  * Uncontrolled symptomatic cardiac arrhythmia,
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Diagnosed to have any of the following condition(s), and/or have undergone any one of the following procedure(s) =< 3 months prior to registration:

  * Symptomatic thrombotic or hemorrhagic cerebral vascular accident
  * Coronary bypass graft
  * Angioplasty
  * Myocardial infarction
* Patients having continuing >= grade 2 adverse events (excluding alopecia) due to agents (chemotherapy or radiotherapy) administered > 4 weeks prior to registration based on Common Terminology Criteria for Adverse Events (CTCAE version 4.0) =< grade 1
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
  * NOTE: because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MK-2206, breastfeeding should be discontinued if the mother is treated with MK-2206; women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* HIV-positive patients on combination antiretroviral therapy; NOTE: HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with MK-2206; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Recent major surgery =< 4 weeks prior to registration (excluding the placement of vascular access), or minor surgery =< 2 weeks prior to registration
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption) that impairs patients ability to swallow MK-2206 tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigette Ma, Principal Investigator — Mayo Clinic
Locations (8):
- United States (4):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong, China
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
  - Johns Hopkins Singapore International Medical Centre, Singapore

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 47 [32 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 19
Region of Enrollment [Number; unit: participants]
  Singapore | 9
  Hong Kong | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Alive and Progression-free
Description: The primary endpoint of this trial is the proportion of patients alive and progression-free at 6 months. Progression status is evaluated using RECIST version 1.1. A Progression is defined as either: At least one new malignant lesion, which also includes any lymph node that was normal at baseline (less than 1.0 cm short axis) and increased to greater than or equal to 1 cm short axis during follow up. Or, at least a 20% increase in sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 21
participants
  Alive and Progression Free | 9
  Dead or Progression | 12

2. Primary Outcome: Confirmed Response Rate Defined to be a CR or PR Noted as the Objective Status on 2 Consecutive Evaluations at Least 4 Weeks Apart
Description: Evaluated using RECIST version 1.1. A Complete Response (CR) requires disappearance of all target lesions and each target lymph node must have reduction in short axis to <1.0 cm. A Partial Response (PR) requires at least a 30% decrease in the sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation. The confirmed response rate is reported as the number of participants with confirmed responses divided by the number of evaluated participants.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 21
percentage of participants
  Complete Response | 0
  Partial Response | 4.8

3. Secondary Outcome: Adverse Events Associated With the Agent Graded Based on CTCAE Version 4.0
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns. Only the severe or worse adverse events will be assessed, regardless of relationship to the study treatment. The number of patients reporting a grade 3 or higher event were counted.
Time Frame: Up to 30 days after completion of study treatment
Population: All patients that began protocol treatment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 21
Participants
  Grade 3+ Adverse Event | 13
  Grade 4+ Adverse Event | 0

4. Secondary Outcome: Overall Survival
Description: Estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, assessed up to 3 years
Population: All patients that started protocol therapy were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 21
months | 10.0 [5.9 to 20.0]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from registration to the time of progression or death, whichever occurs first. Estimated using the method of Kaplan-Meier.
Time Frame: From registration to the first of either death due to any cause or progression, assessed up to 3 years
Population: All patients who began protocol treatment were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 21
months | 3.5 [0.9 to 7.3]

6. Secondary Outcome: Best Response (Complete Response vs Partial Response vs Stable Disease vs Progression)
Description: Evaluated using RECIST version 1.1. A Complete Response (CR) requires disappearance of all target lesions and each target lymph node must have reduction in short axis to <1.0 cm. A Partial Response (PR) requires at least a 30% decrease in the sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation. Progressive Disease (PD) is defined as either a new lesion of a 20% increase in the sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes. Stable Disease (SD) is defined as not having a PD, CR, or PR.
Time Frame: Up to 3 years
Population: All patients who began protocol treatment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 21
Participants
  Stable Disease | 11
  Partial Response (PR) | 1
  Cmplete Response (CR) | 0
  Progressive Disease | 9

7. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented.
Time Frame: The date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented, assessed up to 3 years
Population: Analysis not conducted due to having too few patients with evaluable for this endpoint.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Serious Adverse Events (participants affected / at risk) | 10/21
Other Adverse Events (participants affected / at risk) | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=21)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=21)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2)
Conjunctivitis (Eye disorders) | 4 (5)
Dry eye (Eye disorders) | 1 (3)
Eye disorders - Other, specify (Eye disorders) | 2 (6)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (10)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 9 (34)
Fever (General disorders) | 4 (5)
Flu like symptoms (General disorders) | 1 (5)
Infusion site extravasation (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (2)
Lip infection (Infections and infestations) | 1 (3)
Papulopustular rash (Infections and infestations) | 1 (6)
Skin infection (Infections and infestations) | 1 (2)
Upper respiratory infection (Infections and infestations) | 4 (5)
Alanine aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (9)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (7)
Weight loss (Investigations) | 4 (15)
Anorexia (Metabolism and nutrition disorders) | 4 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Paresthesia (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (6)
Urinary urgency (Renal and urinary disorders) | 1 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (25)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (33)
Flushing (Vascular disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less